CLINICAL TRIAL: NCT00598273
Title: AFX01-11: A Phase 3, Randomized, Active-controlled, Open-label, Multi-center Study of the Safety and Efficacy of Peginesatide for the Correction of Anemia in Patients With Chronic Renal Failure (CRF) Not on Dialysis and Not on Erythropoiesis Stimulating Agent (ESA) Treatment
Brief Title: Safety & Efficacy of Peginesatide for the Treatment of Anemia in Participants With Chronic Renal Failure Not on Dialysis
Acronym: PEARL 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Affymax (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFX01-11
Record Dates: First submitted 2008-01-10; First posted 2008-01-21 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Renal Failure; Chronic Kidney Disease; Anemia
Keywords: anemia; chronic kidney disease; CKD; chronic renal failure; CRF; erythropoietin; EPO; erythropoiesis stimulating agent; ESA; Hematide™; hemoglobin; Hb; Hgb; Omontys; peginesatide; red blood cell; red blood cell production
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Anemia | interventions — peginesatide; hematide; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Peginesatide 0.025 mg/kg (Experimental)
  Interventions: Drug: peginesatide
- Peginesatide 0.04 mg/kg (Experimental)
  Interventions: Drug: peginesatide
- Darbepoetin Alfa (Active Comparator)
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: peginesatide — Participants received peginesatide by subcutaneous injection once every 4 weeks. The starting dose was 0.025 milligram per kilogram (mg/kg) and was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 grams per deciliter (g/dL).
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Peginesatide 0.025 mg/kg
Drug: peginesatide — Participants received peginesatide by subcutaneous injection once every 4 weeks. The starting dose was 0.04 mg/kg and was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 g/dL.
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Peginesatide 0.04 mg/kg
Drug: Darbepoetin alfa — As prescribed, starting dose of 0.75 microgram per kilogram (mcg/kg) administered by subcutaneous injection once every 2 weeks. The dose was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 g/dL.
  Other Names: Aranesp
  Arms: Darbepoetin Alfa

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of peginesatide for the treatment of anemia in participants with chronic kidney disease, who are not on dialysis and not on erythropoiesis stimulating agent (ESA) treatment.

DETAILED DESCRIPTION:
Anemia associated with chronic kidney disease is due to several factors, primarily the inability of the diseased kidneys to produce adequate amounts of endogenous erythropoietin. Ancillary factors include the shortened lifespan of red blood cells, iron and other nutritional deficiencies, infection, and inflammation. The presence and severity of anemia are related to the duration and extent of kidney failure. Anemia is associated with increased mortality, increased likelihood of hospitalization, reduced cognitive function, and increased left ventricular hypertrophy and heart failure.

Erythropoiesis stimulating agents have been established as a treatment for anemia in chronic renal failure subjects, and have improved the management of anemia over alternatives such as transfusion. Peginesatide is a parenteral formulation developed for the treatment of anemia in patients with chronic kidney disease. Peginesatide binds to and activates the human erythropoietin receptor and stimulates erythropoiesis in human red cell precursors in a manner similar to other known erythropoiesis-stimulating agents.

Study participants received doses of peginesatide administered once every 4 weeks or darbepoetin alfa administered once every 2 weeks. Total commitment time for this study was a 4 week screening period followed by a minimum of 52 weeks of study treatment. Eligible participants were randomized in equal proportions to two peginesatide treatment regimens and one control, darbepoetin alfa, treatment regimen.

To evaluate the cardiovascular safety of peginesatide, a cardiovascular composite safety endpoint (CSE) was defined for use in prospectively planned analyses which combined cardiovascular safety data from the four Phase 3 peginesatide studies (NCT00598273, NCT00597753, NCT00598442, and NCT00597584). The CSE consisted of six events: death, stroke, myocardial infarction, and serious adverse events of congestive heart failure, unstable angina, and arrhythmia. An independent Event Review Committee (ERC) was used to provide blinded adjudication of potential CSE events.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic renal failure with an estimated glomerular filtration rate < 60 milliliter per minute per 1.73m^2 and not expected to begin dialysis for at least 12 weeks.
2. Two consecutive hemoglobin values ≥ 8.0 g/dL and < 11.0 g/dL within 4 weeks prior to randomization.

Exclusion Criteria:

1. Females who are pregnant or breast-feeding.
2. Treatment with an ESA in the 12 weeks prior to randomization.
3. Known intolerance to any ESA, parenteral iron supplementation, or pegylated molecule.
4. Prior chronic hemodialysis or chronic peritoneal dialysis treatment.
5. Known bleeding or coagulation disorder.
6. Known hematologic disease or cause of anemia other than renal disease
7. Poorly controlled hypertension
8. Evidence of active malignancy within one year prior to randomization.
9. A scheduled kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President, Clinical Development, Study Director — Affymax
Locations (68):
- United States (65):
  - Research Facility, Montgomery, Alabama
  - Research Facility, Tempe, Arizona
  - Research Facility, Hot Springs, Arkansas
  - Research Facility, Bakersfield, California
  - Research Facility, Chula Vista, California
  - Research Facility, Glendale, California
  - Research Facility, Huntington Beach, California
  - Research Facility, Los Angeles, California
  - Research Facility, Orange, California
  - Research Facility, Paramount, California
  - Research Facility, Pasadena, California
  - Research Facility, Riverside, California
  - Research Facility, San Dimas, California
  - Research Facility, Stanford, California
  - Research Facility, Whittier, California
  - Research Facility, Yuba City, California
  - Research Facility, Thornton, Colorado
  - Research Facility, Washington D.C., District of Columbia
  - Research Facility, Holly Hill, Florida
  - Research Facility, Hudson, Florida
  - Research Facility, Miami, Florida
  - Research Facility, Ocala, Florida
  - Research Facility, Orlando, Florida
  - Research Facility, Tampa, Florida
  - Research Facility, Augusta, Georgia
  - Research Facility, Honolulu, Hawaii
  - Research Facility, Chicago, Illinois
  - Research Facility, Evergreen Park, Illinois
  - Research Facility, Hines, Illinois
  - Research Facility, Evansville, Indiana
  - Research Facility, Lafayette, Indiana
  - Research Facility, Wichita, Kansas
  - Research Facility, Shreveport, Louisiana
  - Research Facility, Bethesda, Maryland
  - Research Facility, Fall River, Massachusetts
  - Research Facility, Worcester, Massachusetts
  - Research Facility, Midland, Michigan
  - Research Facility, Columbus, Mississippi
  - Research Facility, Kansas City, Missouri
  - Research Facility, Northfield, New Jersey
  - Research Facility, Toms River, New Jersey
  - Research Facility, Binghamton, New York
  - Research Facility, Great Neck, New York
  - Research Facility, Mineola, New York
  - Research Facility, Charlotte, North Carolina
  - Research Facility, Oklahoma City, Oklahoma
  - Research Facility, Bend, Oregon
  - Research Facility, Portland, Oregon
  - Research Facility, Allentown, Pennsylvania
  - Research Facility, Erie, Pennsylvania
  - Research Facility, Johnstown, Pennsylvania
  - Research Facility, Providence, Rhode Island
  - Research Facility, Orangeburg, South Carolina
  - Research Facility, Rock Hill, South Carolina
  - Research Facility, Clarksville, Tennessee
  - Research Facility, Knoxville, Tennessee
  - Research Facility, Nashville, Tennessee
  - Research Facility, Austin, Texas
  - Research Facility, Corpus Christi, Texas
  - Research Facility, Corsicana, Texas
  - Research Facility, Edinburg, Texas
  - Research Facility, Houston, Texas
  - Research Facility, San Antonio, Texas
  - Research Facility, Salem, Virginia
  - Research Facility, Bluefield, West Virginia
- Puerto Rico (3):
  - Research Facility, Caguas
  - Research Facility, Ponce
  - Research Facility, San Juan

REFERENCES:
- [Result] Macdougall IC, Provenzano R, Sharma A, Spinowitz BS, Schmidt RJ, Pergola PE, Zabaneh RI, Tong-Starksen S, Mayo MR, Tang H, Polu KR, Duliege AM, Fishbane S; PEARL Study Groups. Peginesatide for anemia in patients with chronic kidney disease not receiving dialysis. N Engl J Med. 2013 Jan 24;368(4):320-32. doi: 10.1056/NEJMoa1203166. PMID 23343062
- [Derived] Fishbane S, Schiller B, Locatelli F, Covic AC, Provenzano R, Wiecek A, Levin NW, Kaplan M, Macdougall IC, Francisco C, Mayo MR, Polu KR, Duliege AM, Besarab A; EMERALD Study Groups. Peginesatide in patients with anemia undergoing hemodialysis. N Engl J Med. 2013 Jan 24;368(4):307-19. doi: 10.1056/NEJMoa1203165. PMID 23343061

RESULTS

PARTICIPANT FLOW:
Groups:
- Peginesatide 0.025 mg/kg: Participants received peginesatide by subcutaneous injection once every 4 weeks. The starting dose was 0.025 milligram per kilogram (mg/kg) and was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 grams per deciliter (g/dL).
- Peginesatide 0.04 mg/kg: Participants received peginesatide by subcutaneous injection once every 4 weeks. The starting dose was 0.04 mg/kg and was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 g/dL.
- Darbepoetin Alfa: Participants received a starting dose of 0.75 microgram per kilogram (mcg/kg) administered by subcutaneous injection once every 2 weeks, as prescribed. The dose was adjusted throughout the study to maintain a hemoglobin target range of 11.0-12.0 g/dL.
Period: Overall Study
Arm/Group | Peginesatide 0.025 mg/kg | Peginesatide 0.04 mg/kg | Darbepoetin Alfa
Started | 161 | 165 | 164
Completed | 120 | 127 | 125
Not Completed | 41 | 38 | 39
Not completed — Adverse Event | 4 | 5 | 2
Not completed — Death | 6 | 12 | 8
Not completed — Lost to Follow-up | 8 | 3 | 5
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 12 | 10 | 10
Not completed — Noncompliance | 3 | 2 | 3
Not completed — Relocation | 0 | 2 | 4
Not completed — Renal transplant | 1 | 0 | 1
Not completed — Site elected to close | 1 | 0 | 0
Not completed — Started dialysis | 6 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peginesatide 0.025 mg/kg | Peginesatide 0.04 mg/kg | Darbepoetin Alfa | Total
Number analyzed (Participants) | 161 | 165 | 164 | 490
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 70 | 63 | 65 | 198
  >=65 years | 91 | 102 | 99 | 292
Age Continuous [Mean (Standard Deviation); unit: years] | 67.1 (13.51) | 67.1 (12.73) | 66.4 (14.25) | 66.9 (13.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 84 | 102 | 279
  Male | 68 | 81 | 62 | 211

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin Between Baseline and the Evaluation Period
Description: The baseline hemoglobin value is defined as the mean of three hemoglobin values: the two most recent hemoglobin values taken prior to the day of randomization and the value obtained on the day of randomization. The mean hemoglobin during the Evaluation Period for each participant is calculated as the mean of the available hemoglobin values during Study Weeks 25 through 36.
Time Frame: Baseline and Weeks 25-36
Population: Full Analysis Population: All randomized participants who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Peginesatide 0.025 mg/kg | Peginesatide 0.04 mg/kg | Darbepoetin Alfa
Number analyzed (Participants) | 161 | 165 | 164
g/dL
  Baseline [N=161, 165, 164] | 10.05 (0.623) | 9.95 (0.685) | 10.05 (0.638)
  Evaluation Period [N=141, 151, 151] | 11.47 (0.731) | 11.61 (0.856) | 11.47 (0.747)
  Change from Baseline [N=141, 151, 151] | 1.39 (0.866) | 1.64 (0.965) | 1.37 (0.861)
Statistical Analysis 1: Comparison: Peginesatide 0.025 mg/kg vs Darbepoetin Alfa; The sample size for this study was determined based on a two-group evaluation of non-inferiority in means with a non-inferiority margin (Δ) of -1.0 g/dL (one-sided significance level of 0.0125, or, comparably, a two-sided significance level of 0.025). A sample size of 450 (150 per treatment group) provided power greater than 99% for the evaluation of non-inferiority, assuming an expected treatment difference of 0.0 g/dL and a pooled standard deviation of 1.5 g/dL; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of -1.0 g/dL was used in the primary efficacy assessments. Non-inferiority was established if the lower limit of the two-sided 97.5% confidence interval for the difference between the means of the primary endpoint (peginesatide minus control ESA) was ≥ -1.0 g/dL; ANOVA; The ANOVA cell means model was used to estimate primary efficacy endpoint within the specified cells formed by the combination of treatment and strata; Least Squares Mean Difference = 0.03, 97.5% CI 2-sided [-0.19 to 0.26], Standard Error of Mean 0.099
Statistical Analysis 2: Comparison: Peginesatide 0.04 mg/kg vs Darbepoetin Alfa; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.26, 97.5% CI 2-sided [0.04 to 0.48], Standard Error of Mean 0.098

2. Secondary Outcome: Proportion of Participants Who Receive Red Blood Cell (RBC) Transfusions During the Correction and Evaluation Periods
Time Frame: Weeks 0 to 36
Population: Full Analysis Population: All randomized participants who received at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Peginesatide 0.025 mg/kg | Peginesatide 0.04 mg/kg | Darbepoetin Alfa
Number analyzed (Participants) | 161 | 165 | 164
percentage of participants | 0.062 | 0.073 | 0.049
Statistical Analysis 1: Comparison: Peginesatide 0.025 mg/kg vs Darbepoetin Alfa; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.25, 95% CI 2-sided [0.51 to 3.10]
Statistical Analysis 2: Comparison: Peginesatide 0.04 mg/kg vs Darbepoetin Alfa; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.48, 95% CI 2-sided [0.62 to 3.56]

3. Secondary Outcome: Proportion of Participants Achieving Hemoglobin Response During the Correction and Evaluation Periods.
Description: A hemoglobin response is defined as hemoglobin increase of ≥ 1.0 gram per deciliter (g/dL) above baseline and a hemoglobin ≥ 11.0 g/dL without RBC transfusion during the previous 8 weeks.
Time Frame: Weeks 0 to 36
Population: Full Analysis Population: All randomized participants who received at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Peginesatide 0.025 mg/kg | Peginesatide 0.04 mg/kg | Darbepoetin Alfa
Number analyzed (Participants) | 161 | 165 | 164
percentage of participants | 0.932 | 0.939 | 0.939
Statistical Analysis 1: Comparison: Peginesatide 0.025 mg/kg vs Darbepoetin Alfa; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.94 to 1.05]
Statistical Analysis 2: Comparison: Peginesatide 0.04 mg/kg vs Darbepoetin Alfa; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.95 to 1.06]

ADVERSE EVENTS:
Arm/Group | Peginesatide 0.025 mg/kg | Peginesatide 0.04 mg/kg | Darbepoetin Alfa
Serious Adverse Events (participants affected / at risk) | 77/161 | 75/165 | 71/164
Other Adverse Events (participants affected / at risk) | 124/161 | 123/165 | 116/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide 0.025 mg/kg (N=161) | Peginesatide 0.04 mg/kg (N=165) | Darbepoetin Alfa (N=164)
Anaemia (Blood and lymphatic system disorders) | 5 | 5 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 15 | 16 | 14
Atrial fibrillation (Cardiac disorders) | 3 | 7 | 3
Myocardial infarction (Cardiac disorders) | 1 | 6 | 4
Acute myocardial infarction (Cardiac disorders) | 4 | 3 | 1
Bradycardia (Cardiac disorders) | 1 | 2 | 4
Coronary artery disease (Cardiac disorders) | 2 | 2 | 3
Angina pectoris (Cardiac disorders) | 2 | 1 | 2
Cardiac arrest (Cardiac disorders) | 2 | 2 | 1
Cardio-respiratory arrest (Cardiac disorders) | 2 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Nodal arrhythmia (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2
Ileus (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 2 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhagic ascites (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 3 | 0 | 3
Asthenia (General disorders) | 2 | 3 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 2
Death (General disorders) | 1 | 1 | 0
Generalised oedema (General disorders) | 1 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Chronic hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 10 | 8 | 9
Urinary tract infection (Infections and infestations) | 5 | 9 | 7
Cellulitis (Infections and infestations) | 6 | 5 | 3
Sepsis (Infections and infestations) | 4 | 1 | 3
Osteomyelitis (Infections and infestations) | 0 | 5 | 1
Bacteraemia (Infections and infestations) | 2 | 1 | 0
Catheter sepsis (Infections and infestations) | 2 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 2
Septic shock (Infections and infestations) | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1
Catheter related infection (Infections and infestations) | 0 | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 1 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0
Carbuncle (Infections and infestations) | 1 | 0 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 1
Endocarditis enterococcal (Infections and infestations) | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1
Fungaemia (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Vulval abscess (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0
Cardiac enzymes increased (Investigations) | 0 | 0 | 1
Electrocardiogram change (Investigations) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 7 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 4 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 5
Fluid overload (Metabolism and nutrition disorders) | 1 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 2 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0
Anoxic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Dementia (Nervous system disorders) | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1 | 0
Syncope vasovagal (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 3 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 21 | 13 | 9
Renal failure chronic (Renal and urinary disorders) | 12 | 3 | 8
Azotaemia (Renal and urinary disorders) | 4 | 3 | 6
Renal failure (Renal and urinary disorders) | 5 | 4 | 4
Haematuria (Renal and urinary disorders) | 1 | 2 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 2
Renal impairment (Renal and urinary disorders) | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 2 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0 | 0
Cystitis erosive (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Neurogenic bladder (Renal and urinary disorders) | 1 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 3 | 5 | 5
Hypertensive crisis (Vascular disorders) | 1 | 1 | 2
Hypotension (Vascular disorders) | 2 | 1 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 2
Aortic aneurysm (Vascular disorders) | 1 | 0 | 1
Hypertensive emergency (Vascular disorders) | 2 | 0 | 0
Malignant hypertension (Vascular disorders) | 1 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0
Intermittent claudication (Vascular disorders) | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Peripheral artery dissection (Vascular disorders) | 0 | 0 | 1
Steal syndrome (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide 0.025 mg/kg (N=161) | Peginesatide 0.04 mg/kg (N=165) | Darbepoetin Alfa (N=164)
Hyperparathyroidism secondary (Endocrine disorders) | 13 | 4 | 6
Nausea (Gastrointestinal disorders) | 27 | 15 | 22
Vomiting (Gastrointestinal disorders) | 23 | 10 | 15
Diarrhoea (Gastrointestinal disorders) | 22 | 17 | 22
Constipation (Gastrointestinal disorders) | 20 | 15 | 16
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 | 11 | 8
Abdominal pain (Gastrointestinal disorders) | 9 | 6 | 4
Oedema peripheral (General disorders) | 31 | 27 | 18
Fatigue (General disorders) | 15 | 7 | 15
Pyrexia (General disorders) | 11 | 6 | 6
Oedema (General disorders) | 7 | 11 | 3
Urinary tract infection (Infections and infestations) | 22 | 24 | 24
Nasopharyngitis (Infections and infestations) | 15 | 18 | 11
Upper respiratory tract infection (Infections and infestations) | 15 | 17 | 15
Bronchitis (Infections and infestations) | 9 | 5 | 7
Cellulitis (Infections and infestations) | 8 | 9 | 3
Influenza (Infections and infestations) | 8 | 9 | 4
Contusion (Injury, poisoning and procedural complications) | 12 | 8 | 6
Fall (Injury, poisoning and procedural complications) | 12 | 15 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 32 | 22 | 27
Hyperphosphataemia (Metabolism and nutrition disorders) | 22 | 8 | 11
Metabolic acidosis (Metabolism and nutrition disorders) | 11 | 7 | 13
Hypoglycaemia (Metabolism and nutrition disorders) | 10 | 8 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 11 | 4
Gout (Metabolism and nutrition disorders) | 7 | 9 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 15 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 19 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 17 | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 | 17 | 17
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 11 | 5
Headache (Nervous system disorders) | 15 | 12 | 13
Dizziness (Nervous system disorders) | 14 | 19 | 24
Insomnia (Psychiatric disorders) | 11 | 8 | 11
Anxiety (Psychiatric disorders) | 9 | 12 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 14 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 14 | 13
Rash (Skin and subcutaneous tissue disorders) | 17 | 9 | 8
Hypertension (Vascular disorders) | 24 | 16 | 17
Hypotension (Vascular disorders) | 7 | 10 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication of the primary safety and efficacy results will include data from all appropriate study sites. Either after the first multicenter publication, or following 36 months after the completion of the study, Investigators are free to publish; such publications may not contain Sponsor Confidential Information and may be subject to Sponsor review 60 days prior to submission for publication.